CLINICAL TRIAL: NCT05137106
Title: Assessment of Effectiveness of Dry Needling for Treating Shoulder Pain: a Randomized Controlled Trial
Brief Title: Assessment of Effectiveness of Dry Needling for Treating Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gran Rosario (Other)
Responsible Party: Principal Investigator, Leonardo Intelangelo, Head of the University Center for Assistance, Teaching and Research, University of Gran Rosario
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: University of Gran Rosario; Reference number 19/17 (Registry Identifier: Ethics Committee for Research in Humans of the Instituto Universitario Italiano de Rosario)
Record Dates: First submitted 2021-11-10; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Chronic Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Active Dry Needling Sham Dry Needling
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participants and Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Dry Needling (Experimental): Active dry needling (ADN). Intramuscular insertion Intervention/treatment. All participants in this group received an ADN session with an intramuscular insertion of a 25 mm X 0.22 mm JEMCO acupuncture needle into the infraspinatus muscle. The dry needling was performed with the rapid entry and exit technique.
  Interventions: Other: Active Dry Needling
- Sham Dry needling (Sham Comparator): Sham dry needling (SDN). All participants in this group received one session of SDN with a 25 mm X 0.22 mm JEMCO acupuncture needle over the infraspinatus region. To ensure that the blunt needles did not puncture the skin during the experimental session (and for patient comfort), each needle was individually cut and polished and checked for sharpness against the investigator's fingertip. As a precaution against infection, each patient was treated with a separate dummy needle.
  Interventions: Other: Sham Dry needling

INTERVENTIONS:
Other: Active Dry Needling — All participants in this group received an ADN session with an intramuscular insertion of a 25 mm X 0.22 mm acupuncture needle into the infraspinatus muscle. The dry needling was performed with the rapid entry and exit technique.
  Arms: Active Dry Needling
Other: Sham Dry needling — All participants in this group received one session of SDN with a 25 mm X 0.22 mm acupuncture needle over the infraspinatus region. To ensure that the blunt needles did not puncture the skin during the experimental session (and for patient comfort), each needle was individually cut and polished and checked for sharpness against the investigator's fingertip. As a precaution against infection, each patient was treated with a separate dummy needle.
  Arms: Sham Dry needling

SUMMARY:
The aim of the study is to evaluate the effects of active dry needling (aDN) in the treatment of myofascial trigger points of the infraspinatus muscle (MTP). For this purpose, this technique was compared to placebo dry needling (pDN) for short-term pain relief and increased glenohumeral internal rotation range. The second objective is to explore whether improvements in perceived pain and functional capacity correlate with changes in electromyographic activity.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled clinical trial comprising a sample of 30 volunteers with unilateral shoulder pain of both sexes, aged 18 to 35 years. They were clinically evaluated to assess inclusion and exclusion criteria. For inclusion in the study, volunteers had unilateral shoulder pain for more than 3 months and were symptomatic at the time of evaluation. The volunteers were randomized into two groups (G1: active dry needling) versus (G2: placebo dry needling). The procedure was performed by one investigator, while outcome measures (pressure pain thresholds, VAS, glenohumeral internal rotation deficit, and muscle activity) were assessed by other investigators, ensuring a double-blinded evaluation of the experiment. Volunteers were recruited through social networks and emails. The study was conducted in two experimental sessions on separate days, at least 48-72 hours apart to avoid carry-over effects. Primary and secondary outcomes were assessed at baseline, immediately after and 48-72 hours after dry needling.

Assessment of infraspinatus and middle deltoid muscle activity was performed by electromyography (EMG). For the EMG protocol, the patient remained standing while holding a distal load, the magnitude of which depended on the patient's weight. In patients weighting less than 68 kg, a load of 1.5 kg was used; those weighting more than 68 kg lifted 2.5 kg. After a brief familiarization period, patients were asked to perform 5 repetitions of shoulder elevation in a scapular plane with external rotation and elbow extended, ranging from 30° to 90°. EMG recordings were taken during the ascent and descent, with a duration of 3 seconds at each stage. The movement was synchronized using a metronome so that there was as little variability as possible between participants.

The study is original and there are no previously published data available. Thus, data obtained from the pilot study were used for sample size calculation. The variable with the lowest coefficient of determination (R-squared) was considered as a primary outcome (pain perceived by visual analog scale), and applied as input for the calculation. The analysis was performed with an effect size of 0.76, an alpha of 5% and a power of 95%. The results indicated that a total of 22 volunteers were needed. Assuming a loss of 20%, each group consists of 14 volunteers (with a total sample of 28 volunteers). The sample calculation was performed using the G-Power 3.1.9.7 software.

The study was pre registered in the brazilian database (www.ensaiosclinicos.gov.br) before starting data collection, although identifier were not provided.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with unilateral shoulder pain
* Glenohumeral internal rotation deficit
* Presence of active myofascial trigger point in the infraspinatus muscle

Exclusion Criteria:

* Previous surgery in the upper limb
* Previous physiotherapy treatments in the shoulder
* Dry needling contraindications
* Previous dry needling experience to mantain the blinding

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain intensity | At baseline, immediately after the intervention, 72 hours after the intervention
  The Visual Analogue Scale (VAS) was used to assess pain intensity. This scale consists of a sequence of numbers from 0 to 10, in which 0 represents "no pain" and 10 represents "worst pain imaginable".

SECONDARY OUTCOMES:
Change in Pressure Pain Threshold | At baseline, immediately after the intervention, 72 hours after the intervention
  Pressure Pain Thresholds (PPT) were quantified bilaterally through a pressure algometer at the medial portion of the infraspinatus muscle and at the medial portion of the deltoid muscle. Three measurements were taken at intervals of 30 seconds and the mean value was recorded. To determine PPT, the pressure was increased at a rate of approximately 1 kg/second. Patients were asked to raise their arm when they perceived the pressure changing to pain, stopping the estimation at this point.
Changes in Range of motion | At baseline, immediately after the intervention, 72 hours after the intervention
  The examiners assessed both shoulder's internal rotation range of motion with an inclinometer.
Changes in EMG activity | At baseline, immediately after the intervention, 72 hours after the intervention
  Electrical activity from infraspinatus and deltoid muscles was recorded using surface electromyography (sEMG). The signal was normalized using the maximal isometric voluntary contraction (MIVC). The sEMG data were collected during a shoulder elevation task. Electrode placement, data collection and processing were performed according to Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles standards.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Gran Rosario, Rosario, Santa Fe Province, Argentina

IPD SHARING:
Plan to Share IPD: Undecided